CLINICAL TRIAL: NCT06439485
Title: Phase I/II Trial of Pemigatinib in Combination With Atezolizumab and Bevacizumab for Treatment of Advanced Cholangiocarcinoma With FGFR2 Fusion
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0106; NCI-2024-04693 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cholangiocarcinoma; FGFR2 Fusion
MeSH Terms: interventions — pemigatinib; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (Experimental): Participants enrolled in Part 1, the dose of pemigatinib the participant receive will depend on when the participant join this study. Up to 2 dose levels of pemigatinib will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the highest dose level of pemigatinib. A second group will receive a lower dose of pemigatinib than the group before it, if intolerable side effects are seen.
  Interventions: Drug: Pemigatinib; Drug: Atezolizumab; Drug: Bevacizumab
- Part 2 (Experimental): Participants in Part 2, you will receive pemigatinib at the recommended dose that was found in Part 1.
  Interventions: Drug: Pemigatinib; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemigatinib — Given by PO
Drug: Atezolizumab — Given by PO and IV
  Other Names: MPDL3280A; TECENTRIQ
Drug: Bevacizumab — Given by PO and IV
  Other Names: Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF

SUMMARY:
To learn if pemigatinib in combination with atezolizumab and bevacizumab can help to control cholangiocarcinoma.

DETAILED DESCRIPTION:
Primary Objectives:

• To assess the antitumor activity of the treatment combinations based on objective response rate (ORR) Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. This assessment will be confirmed in the next scheduled scan.

Secondary Objectives:

1. To determine the safety and recommended phase 2 dose (RP2D) of the triple combination of pemigatinib with bevacizumab and atezolizumab in participants with FGFR-altered metastatic CCA.
2. To evaluate the duration of response in participants with best overall response of complete response (CR) or partial response (PR).
3. To evaluate PFS defined as the time from the start of study treatment to disease progression or death, whichever occurs first.
4. To evaluate the duration of OS defined as the time from the start of study treatment to death from any cause.
5. To evaluate the clinical benefit rate defined as the proportion of participants with best overall response of CR, PR, or stable disease.
6. To evaluate safety and endpoints 2-5 with the doublet of pemigatinib with atezolizumab.

Exploratory Objectives:

• To examine the change of the immune microenvironment on treatment by the combination using a validated immune biomarker panel and end-of-treatment genomic markers using cfDNA to study resistance to pemigatinib and response markers from trial medications.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign informed consent.
* Age ≥18 years.
* Has histologically confirmed metastatic or advanced unresectable cholangiocarcinoma.
* Has disease that is measurable per the RECIST v1.1.
* Has at least one measurable target lesion.
* Has FGFR2 fusion or rearrangement in tumor tissue, as determined by CLIA-validated genomic testing of a tumor tissue specimen (DNA-based or RNA-based).
* Is refractory to, has demonstrated intolerance to, had received, or has refused access to, the 1st line systemic therapy including gemcitabine-based therapy with or without immunotherapy including durvalumab or pembrolizumab. Participants who discontinued available standard therapy due to toxicity must have continued evidence of measurable disease.
* Has available a formalin-fixed, paraffin-embedded primary tumor sample.
* Is able to take oral medication and to comply with protocol procedures and scheduled visits..
* Has Eastern Cooperative Oncology Group performance status of 0 or 1
* Has adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1000/µL) without granulocyte colony-stimulating factor support
* Platelet count ≥ 100 × 109/L (100,000/µL) without transfusion
* Hemoglobin ≥ 90 g/L (9 g/dL), participants may be transfused to meet this criterion.
* Aspartate amino transferate (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × upper limit of normal (ULN), with the following exceptions:
* Participants with documented liver metastases: AST and ALT ≤ 5 × ULN
* Participants with documented liver or bone metastases: ALP ≤ 5 × ULN
* Serum bilirubin ≤ 1.5 × ULN with the following exception:
* Participants with known Gilbert disease: serum bilirubin ≤ 3 × ULN
* Serum creatinine ≤ 1.5 × ULN
* Serum albumin ≥ 25 g/L (2.5 g/dL)
* For participants not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. For patients on anticoagulation, those on therapeutic anticoagulation over 2 weeks are eligible.
* Has a negative human immunodeficiency virus (HIV) test at screening with the following exception: participants with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200 and have an undetectable viral load.
* Has a negative hepatitis B surface antigen (HBsAg) test at screening (unless participant has chronic HBV on anti-viral therapy)
* Has a negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening (unless patient has chronic HBV on anti-viral therapy)
* The HBV DNA test will be performed only for participant who have a negative HBsAg test and a positive total HBcAb test.
* Participants with chronic HBV on antiviral therapy or HCV participants who have completed curative anti-viral therapy can be included.
* Contraception requirements for marketed Roche IMPs or NIMPs should be based on recommendations in the Summary of Product Characteristics or, if there is no Summary of Product Characteristics, national prescribing information. Length of time required for abstinence or use of contraceptives should take into account the reproductive toxicity profile, including genotoxicity and teratogenicity, the size of the molecule, and the number of doses. In the absence of specific delayed-toxicity concerns or safety hypotheses, the following guidelines should be used: Single-dose studies Small Molecules: 5 elimination half-lives or 14 days after the last dose, whichever is longer Large Molecules: 2 elimination half-lives or 28 days after the last dose, whichever is longer Multiple-dose studies Small Molecules: 5 elimination half-lives or 28 days after the last dose, whichever is longer Large Molecules: 2 elimination half-lives or 28 days after the last dose, whichever is longer Options for female contraception are based on the Clinical Trial Facilitation Group "Recommendations related to contraception and pregnancy testing in clinical trials." Three options for female contraception are shown below.
* For women of childbearing potential: agrees to remain abstinent (refrain from heterosexual intercourse) or to use contraceptive methods, and agrees to refrain from donating eggs, as defined below:
* Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of atezolizumab/pemigatinib/bevacizumab. Women must refrain from donating eggs during this same period.
* A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/ or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
* Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. Options for contraception in male patients with pregnant female partners and/ or with female partners of childbearing potential are based on the Clinical Trial Facilitation Group "Recommendations related to contraception and pregnancy testing in clinical trials" and the Roche White Paper regarding contraception for males in clinical trials. Atezolizumab does not require male contraception or condom use; guidelines below apply to other protocol-mandated study treatments.
* For men: agrees to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agrees to refrain from donating sperm, as defined below:
* With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of atezolizumab/pemigatinib/ bevacizumab to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of preventing drug exposure.

Exclusion Criteria:

* Received prior chemotherapy, biologic therapy, immunotherapy, or investigational agent within 3 weeks prior to initiation of study medications.
* Had previous treatment with selective FGFR inhibitors including erdafitinib, infigratinib, or futibatinib.
* Had prior therapy with any VEGFR-targeting agent targeting including bevacizumab, ramucirumab, pazopanib, lenvatinib, and other anti-angiogenesis inhibitors.
* Has a history and/or has current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, vascular system, and lung. Exceptions include calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcifications-these are allowed.
* Has corneal or retinal disorder/keratopathy with current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/ band keratopathy, inflammation, or ulceration, keratoconjunctivitis, or diabetic retinopathy, confirmed by ophthalmic physician. Participants with asymptomatic ophthalmic conditions assessed by the investigator to pose minimal risk for study participation may be enrolled in the study.
* Are currently receiving or are planning to receive during participation in this study, treatment with any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug. Moderate CYP3A4 inhibitors are not prohibited but should be avoided. Medications that increase serum phosphorus and/or calcium concentration are prohibited. Medications associated with hyperphosphatemia and/or hypercalcemia adverse events are searchable in the Leximcomp Online Pharmacy & Formulary available on the Inside MD Anderson Clinical Tools SharePoint site. Participants are not permitted to receive enzyme-inducing anti-epileptic drugs, including carbamazepine, phenytoin, phenobarbital, and primidone.
* Have consumed grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges or products containing juice of these fruits within 7 days prior to first dose of study drug.
* Had a Grade 3-4 gastrointestinal bleed within 3 months prior to enrollment.
* Has a history of deep vein thrombosis, pulmonary embolism, or any other thromboembolism, including portal venous thrombosis within 3 months prior to enrollment. Venous port or catheter thrombosis, incidental asymptomatic pulmonary embolism diagnosed on imaging studies, or superficial venous thrombosis are not considered significant and are allowed.
* Has current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants (including direct oral anticoagulants); thrombolytic agents for therapeutic (as opposed to prophylactic) purpose; use of aspirin (> 325 mg/day); or use of clopidogrel (> 75 mg/day). Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the INR and/or aPTT is within therapeutic limits (according to institution standards) within 7 days prior to initiation of study treatment and the patient has been on a stable dose of anticoagulants for ≥ 2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran and rivaroxaban is not recommended due to bleeding risk.
* Had significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, transient ischemic attack or cerebrovascular accident); unstable arrhythmia; or unstable angina significant cardiovascular disease within 6 months prior to enrollment.
* Has a history of uncontrolled or poorly-controlled hypertension (>150 mmHg systolic or >100 mmHg diastolic).
* Has a history of hypertensive crisis or hypertensive encephalopathy.
* Had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* Has undergone major surgery (including open biopsy, surgical resection, wound revision; or any other major surgery involving entry into a body cavity); or significant traumatic injury within 28 days prior to enrollment; or subcutaneous venous-access-device placement within 7 days prior to enrollment; or anticipates need for major surgical procedure, core biopsy, or other minor surgical procedures during the course of the study. o Note: Placement of a vascular access device should be at least 2 days prior to initiation of study treatment.
* Is receiving chronic antiplatelet therapy, nonsteroidal anti-inflammatory drugs (e.g., ibuprofen, naproxen), dipyridamole, clopidogrel, or similar agents. Once-daily aspirin use (≤325 mg/day) is allowed.
* Has had significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization.
* Has a history of central nervous system disease or evidence of this disease upon physical or neurological examination.
* Has a history of Grade ≥ 2 hemoptysis (defined as ≥ 2.5 mL of bright red blood per episode) within 1 month prior to screening.
* Has a history or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation).
* Has a history of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess, or active GI bleeding within 6 months prior to randomization.
* Has a history of leptomeningeal disease.
* Has uncontrolled tumor-related pain.
* Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Participants should have recovered from the effects of radiation. There is no required minimum recovery period.
* Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy, if appropriate, prior to enrollment.
* Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (at a frequency of at least once monthly) o Participants with indwelling catheters (e.g., PleurX®) are allowed. Has uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL, or corrected serum calcium > ULN).
* Has current evidence of endocrine alterations of calcium/phosphate homeostasis, eg, parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis, and other disorders.
* Has elevated phosphorus or abnormal serum calcium, or phosphorus, or calcium-phosphorus product ≥ 55 mg2/dL2:
* Inorganic phosphorus > 1.02 × ULN Has active or a history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 9 for full list), with the following exceptions:
* Participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study. Participants with controlled Type 1 diabetes mellitus (as determined by the treating physician) who are on an insulin regimen are eligible for the study.
* Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover < 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids • No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet-A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* Has a history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis; or has evidence of active pneumonitis upon screening via computed tomography (CT) scan of the chest.
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Has active tuberculosis.
* Had a major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipates need for a major surgical procedure during the study.
* Had a history of malignancy other than cholangiocarcinoma within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* Had a severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Received treatment with therapeutic oral- or IV antibiotics within 2 weeks prior to initiation of study treatment.
* Participants receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Had a prior allogeneic stem cell or solid organ transplantation • Has any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that may render the patient at high risk from treatment complications.
* Received treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipates need for such a vaccine during treatment or within 5 months after the final dose of treatment. Receipt of SARS-CoV vaccine is allowed.
* Received treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:
* Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
* Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Received treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, or anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipates a need for systemic immunosuppressive medication during study treatment, with the following exceptions:
* Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.
* Participants who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Has a history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Has a known hypersensitivity to Chinese hamster ovary-cell products or to any component of the atezolizumab formulation.
* Has a known allergy or hypersensitivity to any component of the pemigatinib, bevacizumab, or atezolizumab formulations.
* Is pregnant or breastfeeding or intends to become pregnant during study treatment or within 6 months after the final dose of study treatment.
* Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.
* Has a history of hypovitaminosis D requiring supraphysiologic doses (eg, 50,000 UI/weekly) to replenish the deficiency. Vitamin D supplements are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2028-02-22 (Estimated); Study Completion 2030-02-22 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sunyoung Lee, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org